CLINICAL TRIAL: NCT04930289
Title: Global Utilization and Registry Database for Improved Preservation of Donor Lungs
Acronym: GUARDIANLUNG
Status: Enrolling by invitation | Type: Observational
Sponsor: Paragonix Technologies (Industry)
Responsible Party: Sponsor
Other Study IDs: PGX-004
Record Dates: First submitted 2021-06-09; First posted 2021-06-18 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Interstitial Lung Disease; COPD; Cystic Fibrosis; Pulmonary Fibrosis; Pulmonary Arterial Hypertension; Emphysema
MeSH Terms: conditions — Lung Diseases, Interstitial; Pulmonary Disease, Chronic Obstructive; Cystic Fibrosis; Pulmonary Fibrosis; Pulmonary Arterial Hypertension; Emphysema

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (3):
- LungGuard patients: Patients whose donor lung(s) was transported with the LungGuard device.
  Interventions: Device: LungGuard
- Standard Transport Patients: Patients whose donor lung(s) was transported with a method other than the LungGuard
- BAROGuard Patients: Patients whose donor lung(s) was transported with the BAROGuard device.
  Interventions: Device: BAROGuard

INTERVENTIONS:
Device: LungGuard — The LUNGguard is an FDA cleared and is a CE-marked medical device intended to be used for the static hypothermic preservation of lungs during transportation and eventual transplantation into a recipient using cold storage solutions indicated for use with the lungs. The intended organ storage time for the LUNGguard is up to 8 hours.
  Groups: LungGuard patients
Device: BAROGuard — The BAROguard (the "System") is ultraportable hypothermic preservation and transport system intended for use with donor lungs. BAROguard is a legally marketed, FDA cleared medical device in the United States. The intended organ storage time for BAROguard™ is up to 8 hours.
  Groups: BAROGuard Patients

SUMMARY:
The objective of this registry is to collect and evaluate various clinical effectiveness parameters in patients with transplanted donor lung that were preserved and transported within the LUNGguard system, as well as retrospective standard of care patients

DETAILED DESCRIPTION:
GUARDIAN-Lung is a post-market, observational registry of adult and pediatric lung transplant recipient patients whose donor lungs was preserved and transported within the LUNGguard. The data is being collected retrospectively from medical records of patients already transplanted before the initiation of the registry and any new patients who meet the eligibility criteria.

About 500 male and female subjects (including pediatric patients) meeting the study inclusion and exclusion criteria will be enrolled into the study at about 5 clinical sites.

Candidates that fit the eligibility criteria and have had their donor lungs transported with a Paragonix product or a standard of care method can be enrolled. The baseline characteristics and outcomes of the two groups will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Donor and donor lungs matched to the prospective recipient based upon institutional medical practice
* Registered male or female primary lung transplant candidates including pediatric candidates

Exclusion Criteria:

* Donor and donor lungs that do not meet institutional clinical requirements for transplantation
* Patients who are incarcerated persons (prisoners)
* Patients who have had a previous major organ transplant (heart, lungs, liver, kidney, pancreas)
* Patients who are receiving multiple organ transplants

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Primary lung transplant candidates at centers that use the LungGuard device
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2021-10-15 (Actual); Primary Completion 2028-06-15 (Estimated); Study Completion 2029-12-30 (Estimated)

PRIMARY OUTCOMES:
Number of subjects with Primary Graft Dysfunction (PGD) | Post-transplant through 1 year post
  The number of subjects that develop PGD after transplant
Number of subjects with rejection | Post-transplant through 1 year post
  Subjects that show signs to rejection after transplant
Survival | Post-transplant through 1 year post
  patient survival post-transplant
ICU Length of Stay | Transplant through 1 year post-transplant
  Days the subject spent the ICU post-transplant
Hospital Length of Stay | Transplant through 1 year post-transplant
  Days the subject was in the hospital in total after transplant

SECONDARY OUTCOMES:
Number of rehospitalizations | post-transplant through 1 year
  The number of times the subject was readmitted to the hospital after discharged post-transplant
How long subjects needed mechanical support | pre-transplant through 48 hours post-transplant
  Amount of time (minutes) mechanical support (EMCO and ventilator) was needed pre and post transplant

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Hartwig, MD, Principal Investigator — Duke University
Locations (15):
- United States (14):
  - St. Joseph's Hospital and Medical Center, Phoenix, Arizona
  - University of California, San Francisco, San Francisco, California
  - Stanford Medicine, Stanford, California
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - Johns Hopkins University, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Montefiore Hospital, The Bronx, New York
  - Duke Lung Transplant Clinic, Durham, North Carolina
  - Temple University Hospital, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Baylor Scott & White Research Institute, Dallas, Texas
  - The University of Texas Southwestern Medical Center, Dallas, Texas
  - Houston Methodist Hospital, Houston, Texas
  - University of Virginia, Charlottesville, Virginia
- University Hospitals Leuven, Leuven, Belgium